CLINICAL TRIAL: NCT02526589
Title: Does Bloody Urine Predict Urethrovesical Anastomosis Leakage After Radical Prostatectomy
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: R15042
Record Dates: First submitted 2015-08-10; First posted 2015-08-18 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Prostatic Neoplasm; Anastomosis
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Traditionally the watertightness of urethrovesical anastomosis after robotic radical prostatectomy is controlled by cystogram. However, clinical observations and one previous study showed that patients with anastomotic leakage have red coloured urine. If the investigators can verify this finding, the most of the cystograms can be avoided. In this study the investigators estimate urine colour after cystogram and take a picture from urine collecting pag. Later on the pictures are digitally analyzed and compared to cystogram finding.

ELIGIBILITY:
Inclusion Criteria:

* Previous robotic radical prostatectomy
* Catheter removal visit

Exclusion Criteria:

* No urine in urinary collecting bag

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Robotic assisted laparoscopic radical prostatectomy patients. Catheter removal visit.
Sampling Method: Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2015-08; Primary Completion 2017-09-20 (Actual); Study Completion 2017-09-20 (Actual)

PRIMARY OUTCOMES:
Urine colour | 1 week
  correlation of urine colour to cystogram finding

CONTACTS AND LOCATIONS:
Overall Officials: Jarno Riikonen, MD, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No